CLINICAL TRIAL: NCT05527522
Title: Prognostic and Clinical Impact of a Nutritional Intervention in Patients With Chronic Heart Failure
Brief Title: Nutritional Intervention in Malnourished Patients With Chronic Heart Failure
Acronym: PACMAN-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carolina Ortiz Cortes, Doctor, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3/2018
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure; Malnutrition
Keywords: Malnutrition; Heart failure; Nutritional intervention
MeSH Terms: conditions — Heart Failure; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Control arm: Who received the usual practice.
  Interventions: Other: standard practice
- Intervention (Experimental): Intervention arm: Who received an individualized diet, educational intervention with/without nutritional supplements depending on the degree of malnutrition plus usual practice
  Interventions: Combination Product: nutritional and educational intervention; Other: standard practice

INTERVENTIONS:
Combination Product: nutritional and educational intervention — individualized diet plus educational intervention with/without nutritional supplements
  Arms: Intervention
Other: standard practice — The patients received the usual treatment and clinical practice

SUMMARY:
Malnutrition is common in patients with heart failure (HF) and is associated with a worse prognosis.

However, there is little information on the impact of nutritional intervention in malnourished patients with heart failure. Therefore, the aim of our study is to evaluate whether a specific nutritional intervention has an impact on mortality and hospitalizations, quality of life, nutritional status, and functional capacity in patient with heart failure and malnutrition.

DETAILED DESCRIPTION:
A high prevalence of malnutrition has been reported in hospitalized patients with acute heart failure and some studies suggest that personalized treatments or interventions on nutritional status could improve prognosis in these patients. Previous studies have shown that malnutrition is an independent factor associated with worse prognosis not only in hospitalized patients with decompensated HF but also in patients with chronic stable HF. In this sense, it has been postulated that nutritional intervention in malnourished patients with HF could have some prognostic benefit. However, there are very few data published in the literature that have assessed the nutritional status and the benefit of a nutritional intervention in stable ambulatory patients with chronic HF.

Therefore, the aim of this study was to evaluate whether the application of an educational and nutritional intervention in malnourished patients with heart failure improves prognosis, nutritional status, functional capacity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with a confirmed diagnosis of HF according to current criteria established by clinical practice guidelines and who present left ventricular dysfunction documented by echocardiography (LVEF less than 40%).
* Patients with clinical stability in the last 6 months defined as no admissions or decompensations in the last 6 months.
* Patients with malnutrition or at risk of malnutrition according to criteria established by the Mini Nutritional Assessment score (see attached).
* Patients who agree to participate in the study by signing the written informed consent after receiving verbal and written information about the study.

Exclusion Criteria:

* *Dementia or severe cognitive impairment.

  * Dialysis.
  * Already receiving nutritional supplements.
  * Known concomitant oncologic process or other concomitant disease with life expectancy of less than 1 year.
  * Pregnant women.
  * Participation in another clinical trial concurrently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Time to the First Event of Adjudicated Cardiovascular (CV) Death or Adjudicated Hospitalisation for Heart Failure (HHF) | From randomisation until completion 365 days
  [ Time to the first event of adjudicated cardiovascular (CV) death or adjudicated hospitalisation for heart failure (HHF). The incidence rate per 100 patient years (100 * number of patients with event /time at risk [years]) is presented. With time at risk [year] calculated as: Sum of time at risk [days] over all patients in a treatment group / 365.25.
  Patients without a specific endpoint event were censored at the last date the patient was known to be free of the event or at the end of the planned treatment period, whichever was earlier.
  Unit of Measure: Patients with events per 100 patient-years (pt-yrs) at risk.

SECONDARY OUTCOMES:
To assess the impact of the intervention on nutritional status. | baseline and 52 weeks
  Nutritional status will be established according to the Mini Nutritional Assesment (MNA) score, which includes 18 items divided into 4 groups: anthropometry, general condition, dietary aspects and subjective assessment. The nutritional status is classified into 3 groups according to the score obtained: well nourished (equal to or greater than 24 points), at risk of malnutrition (17-23.5 points) and malnourished (less than 17 points), and other biochemical and anthropometric parameters will be collected to complete the nutritional study
To assess the impact of the intervention on quality of life | baseline and 52 weeks. Assessed at baseline, week 12, week 26 and week 52
  Change From Baseline in KCCQ (Kansas City Cardiomyopathy Questionnaire) Clinical Summary Score at Week 52.
  The KCCQ is a 23-item self-administered questionnaire designed to evaluate physical limitations, symptoms (frequency, severity, and changes over time), social limitations, selfefficacy, and quality of life in patients with Heart Failure. The KCCQ-clinical summary score comprises the following domains: Symptom frequency, symptom burden and physical limitation. The score is calculated by summing domain responses and then transforming scores to a 0-100 unit scale with higher scores indicating better health status.
  For patients who died, a worst score (score of 0) is imputed at all subsequent scheduled visits after the date of death.
To assess the impact of the intervention on be assessed by means of the 6-minute test. | baseline and 52 weeks. Assessed at baseline, week 12, week 26 and week 52
  Functional capacity is assessed with the 6-minute test. It consists of measuring the maximum distance that the patient is able to walk in 6 minutes, in a short corridor, simultaneously evaluating the heart rate, oxygen saturation and the degree of dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Ortiz Cortés, Principal Investigator — Carolina Ortiz Cortés
Locations (1):
- Hospital San Pedro de Alcántara, Cáceres, Spain

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT05527522/SAP_000.pdf